CLINICAL TRIAL: NCT00029679
Title: Borage Oil and Ginkgo Biloba (EGb 761) in Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01AT000637-02 (NIH)
Record Dates: First submitted 2002-01-18; First posted 2002-01-21 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Ginkgo Extract; borage oil

INTERVENTIONS:
Drug: Gingko biloba
Drug: Borage oil

SUMMARY:
This study will assess clinical efficacy and/or adverse effects of dietary borage oil (which contains gamma-linolenic acid [GLA]) and Ginkgo biloba in patients with mild persistent to moderate asthma.

DETAILED DESCRIPTION:
The concept of asthma as a condition in which acute and chronic inflammatory changes in airways play a fundamental role is well established. The role of leukotrienes as a crucial element of these inflammatory processes is supported by abundant laboratory and clinical evidence. There is a potential for herbal medicinal approaches to ameliorate leukotriene-mediated inflammation in asthma based on data from the literature and our laboratory. Studies suggest that dietary GLA, found in borage and evening primrose oils, is unique among the (n-6) polyunsaturated fatty acid family members (linolenic acid, GLA and arachidonic acid) in its potential to attenuate inflammatory processes. For instance, there are randomized, placebo-controlled trials (RCT) demonstrating efficacy of dietary GLA in treating patients with rheumatoid arthritis and active synovitis. Ginkgo biloba, a flavonoid-rich extract of leaves of the Ginkgo biloba tree, has been studied in one RCT with asthma patients and is recommended by complementary and alternative practitioners as treatment for allergic inflammation and asthma. Ginkgo biloba supplements have no known adverse effects.

We will assess clinical efficacies and/or adverse effects of dietary borage oil and Ginkgo biloba in patients with asthma in a 17 month RCT. We also propose to delineate whether or not the clinical course of treatment correlates with suppression of leukotriene B4 (LTB4), LTC4 and LTD4 generated by activated polymorphonuclear cells. Additionally, in the Ginkgo biloba arms of study, the in vitro/ex vivo inhibition of histamine release will be assayed, since one of its major constituents, quercetin, is known to be structurally related to cromolyn sodium and has been shown in vitro studies to exhibit similar activities. Furthermore, anti-inflammatory activities of Ginkgo biloba will be compared to those of some of its individual constituents in a series of in vitro experiments. It is hoped that findings from these studies will evolve relatively non-toxic therapeutic alternatives for attenuating bronchial hyperresponsiveness and inflammation in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms (cough, wheeze, chest tightness) consistent with the National Asthma Education Program (NAEP) guidelines for mild persistent to moderate asthma

Exclusion Criteria:

* Severe asthma or mild intermittent asthma by NAEP revised guidelines
* History of vasovagal reactions (nausea, dizziness, flushed/warm) upon having blood drawn
* Pregnancy or lactation
* History of emergency room care in the last 6 months
* History of hospitalization
* Use of prednisone in the past 3 months
* Concurrent pulmonary disease: pulmonary hypertension, cystic fibrosis, sarcoidosis, bronchiectasis, hypersensitivity pneumonitis, restrictive lung disease
* Cigarette smoking within the past 1 year; over 10-pack year history of cigarette smoking in ex-smokers
* Recent (within one month) upper or lower respiratory tract infection

  * The following concurrent medical diagnoses: alcoholism, coronary artery disease, diabetes, HIV infection, chronic hepatitis, uncontrolled hypertension, or a psychiatric disorder that is judged to make full participation difficult
* Use of prednisone in the past 3 months; current use of zileuton (leukotriene receptor antagonists are allowed) or theophylline
* Use of dietary supplements (except for standard dose multiple vitamins such as One-a-day or Centrum) including herbal supplements, mega dose of multiple vitamins/antioxidants, magnesium, fish oil, borage oil, evening primrose oil, black currant oil, fungal oil, G. biloba, quercetin, or mega intake of garlic or onion (subjects will be asked to stop such therapies as a requirement of enrollment)
* Ongoing use of homeopathic remedies or acupuncture, acupressure, therapeutic massage (subjects will be asked to stop such therapies as a requirement of enrollment)

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280
Dates: Start 2000-09; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States